CLINICAL TRIAL: NCT00426621
Title: A 12-Week, Randomized, Double-Blind, Multi-Center, Vehicle-Controlled, Parallel Group Study to Assess the Efficacy and Safety of the Diclofenac Sodium Gel 1% for the Relief of Signs and Symptoms in Patients With Osteoarthritis of the Knee.
Brief Title: Efficacy and Safety of Diclofenac Sodium Gel (DSG) in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Roy Altman, University of California, in Los Angeles, Division of Rheumatology,
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VOSG-PN-316
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: Knee osteoarthritis, degenerative joint disease, knee pain, joint pain, topical NSAID,; diclofenac sodium
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Diclofenac Sodium Gel
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Sodium Gel — 4 grams per knee, 4 times per day, for 12 weeks
  Arms: 1
Drug: Placebo — 4 grams per knee, 4 times per day, for 12 weeks
  Arms: 2

SUMMARY:
This study will test the efficacy and safety of topical diclofenac sodium gel in the treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee

Exclusion Criteria:

* Other rheumatic disease, such as rheumatoid arthritis
* Active gastrointestinal ulcer during the last year
* Known allergy to analgesic drugs
* Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2006-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
pain in the target knee (WOMAC pain index);
functional capacity in the target knee (WOMAC function index); and
global rating of benefit (100 mm Visual Analogue Scale, VAS).

SECONDARY OUTCOMES:
Efficacy of Diclofenac Sodium Gel 1% with regard attainment of:
Low pain intensity in either knee; and
Low functional impairment in either knee.
Safety of Diclofenac Sodium Gel 1% assessed by:
monitoring adverse events; and
laboratory evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Altman, MD, Principal Investigator — University of California, in Los Angeles, Division of Rheumatology, 310 206 7866
Locations (64):
- United States (64):
  - Coastal Clinical Research Inc, Mobile, Alabama
  - River Region Research, LLC, Tallassee, Alabama
  - East Valley Family Physicians, Chandler, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Heartland Research Associates LLC, Arkansas City, Arkansas
  - Lovelace Scientific Research, Inc., Beverly Hills, California
  - MED Investigations, Carmichael, California
  - MED Investigations, Inc., Fair Oaks, California
  - Universal BioPharma Research, Inc., Fresno, California
  - Santa Barbara Clinical Research, Inc, Santa Barbara, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Clinical Research Consultants, LLC, Stratford, Connecticut
  - Seidman Clinical Trials, Delray Beach, Florida
  - Florida Medical Research Institute, Gainesville, Florida
  - South Florida Clinical Research Center, Hollywood, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Suncoast Internal Medicine Consultants, Largo, Florida
  - AppleMed Research, Inc., Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Sunshine Research Center, LLC, Opa-locka, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Andres Patron DO PA, Pembroke Pines, Florida
  - Radiant Research - St Petersburg, Pinellas Park, Florida
  - Sunrise Medical Research, Plantation, Florida
  - Coastal Medical Research, Port Orange, Florida
  - Radiant Research, Stuart, Florida
  - Intermountain Orthopaedics, Boise, Idaho
  - Medical Specialists Clinical Research Center, Munster, Indiana
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Best Clinical Trial, LLC, New Orleans, Louisiana
  - Peter A. Holt, MD, Baltimore, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Phase III Clinical Research, Fall River, Massachusetts
  - Professional Clinical Research, Inc, Cadillac, Michigan
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Internal Medical Associates, Grand Island, Nebraska
  - South Jersey Medical Associates, PA, Blackwood, New Jersey
  - North Carolina Arthritis & Allergy Care Center, Raleigh, North Carolina
  - Rapid Medical Research, Inc, Cleveland, Ohio
  - Radiant Research, Columbus, Ohio
  - Radiant Research, Inc. - Akron, Mogadore, Ohio
  - Clinical Research Source, Inc, Perrysburg, Ohio
  - Neshaminy Medical, PC, Bensalem, Pennsylvania
  - Westminster Family Medicine, Erie, Pennsylvania
  - Feasterville Family Health Care Center, Feasterville, Pennsylvania
  - Southeastern Pennsylvania Medical Institute, Havertown, Pennsylvania
  - Radiant Research, Philadelphia, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research - Anderson, Anderson, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Walter F. Chase, M.D., P.A., Austin, Texas
  - Radiant Research Dallas North, Dallas, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Radiant Research - San Antonio, San Antonio, Texas
  - Texas Research Center, LLP, Sugar Land, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - The Physicians Clinic of Spokane, Spokane, Washington
  - Advanced Healthcare, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Baraf HS, Gloth FM, Barthel HR, Gold MS, Altman RD. Safety and efficacy of topical diclofenac sodium gel for knee osteoarthritis in elderly and younger patients: pooled data from three randomized, double-blind, parallel-group, placebo-controlled, multicentre trials. Drugs Aging. 2011 Jan 1;28(1):27-40. doi: 10.2165/11584880-000000000-00000. PMID 21174485